CLINICAL TRIAL: NCT07088783
Title: The Effect of Mobile Application-Based Education Developed According to Orem's Self-Care Model on Enhancing Self-Care Agency in Patients With Multiple Myeloma: A Randomized Controlled Trial
Brief Title: Mobile App Education Based on Orem's Self-Care Model in Multiple Myeloma Patients
Acronym: OCARE-MM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ozlem (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Sponsor-Investigator, Ozlem, Professor, Faculty of Nursing, Dokuz Eylul University, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DEU-MM-RCT-2024-0923; 2024/09-23 (Other: Dokuz Eylul University Ethics Committee); TDK-2025-3605 (Other: Dokuz Eylul University Scientific Research Projects Coordination Unit (BAP))
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma (MM); Self-care; Quality of Life
Keywords: Multiple Myeloma; Orem's Self-Care Model; Mobile Health Education; Quality of Life; Self-Care Agency
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Two-group parallel design. Participants were randomly assigned to either the intervention group, which received a mobile application-based educational program for 24 weeks, or the control group, which received routine care and a standard brochure.
Who Masked: Participant
Masking Description: Participants were blinded to their group assignment. The investigator was aware of group allocation, as the study is a doctoral thesis project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A mobile application was provided to support self-care and quality of life, based on Orem's Self-Care Deficit Model. Patients were asked to use it regularly for 24 weeks.
  Interventions: Behavioral: Mobile App Education
- Control Group (No Intervention): Participants received routine care and a one-page standard information brochure for cancer patients.

INTERVENTIONS:
Behavioral: Mobile App Education — A 24-week self-care education delivered via a mobile application based on Orem's Self-Care Model
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aims to assess the effectiveness of a mobile application-based education program, developed according to Orem's Self-Care Model, in improving self-care agency and quality of life among patients with multiple myeloma in Turkey. Participants are recruited from the outpatient clinic of a hospital and randomly assigned to either the intervention or control group. The intervention group uses the mobile application for 24 weeks, while the control group continues with routine care and receives a standard one-page brochure commonly distributed to cancer patients. All participants complete a demographic form, the EORTC QLQ-C30, QLQ-MY20, and the Self-Care Agency Scale at baseline, week 12, and week 24. The collected data will be used to compare changes in self-care agency and quality of life between the two groups over time.

DETAILED DESCRIPTION:
This study was conducted to address the self-care needs of patients diagnosed with multiple myeloma, a chronic and complex hematologic cancer. Based on Orem's Self-Care Deficit Nursing Theory, a mobile application was developed to improve patients' self-care agency and quality of life. The intervention group uses the mobile application for 24 weeks, which includes educational content, self-monitoring features, and motivational messages. The control group receives routine care, which includes standard medical follow-up and a one-page general information brochure commonly provided to cancer patients at the hospital. Self-care agency and quality of life are assessed using the Self-Care Agency Scale, EORTC QLQ-C30, and EORTC QLQ-MY20 at three time points: baseline, week 12, and week 24. The results are expected to contribute to evidence-based self-care interventions for patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple myeloma and received at least one course of treatment
* Age 18 or older
* Able to speak and read Turkish
* ECOG performance status of I, II, or III
* Has used at least one Android-based digital tool (e.g., sending text messages, email, using mobile apps)
* Literate (able to read and write)
* Willing to participate and able to provide written informed consent

Exclusion Criteria:

* Not currently diagnosed with multiple myeloma
* Has cognitive or psychological disorders that prevent completing questionnaires or using the mobile application
* Unable to speak or understand Turkish
* Unwilling or unable to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Care Agency Score | Baseline, 12th week, and 24th week
  Self-care agency was assessed using the Self-Care Agency Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to ethical constraints and participant confidentiality concerns in accordance with institutional review board (IRB) approval.

REFERENCES:
- [Background] Hartweg DL, Metcalfe SA. Orem's Self-Care Deficit Nursing Theory: Relevance and Need for Refinement. Nurs Sci Q. 2022 Jan;35(1):70-76. doi: 10.1177/08943184211051369. PMID 34939484
- [Background] Kayser L, Kushniruk A, Osborne RH, Norgaard O, Turner P. Enhancing the Effectiveness of Consumer-Focused Health Information Technology Systems Through eHealth Literacy: A Framework for Understanding Users' Needs. JMIR Hum Factors. 2015 May 20;2(1):e9. doi: 10.2196/humanfactors.3696. PMID 27025228